CLINICAL TRIAL: NCT03420560
Title: A Warmer Room-temperature at 27-28 Centi-degree Will Decrease Propofol Injection Pain
Brief Title: A Warmer Temperature Decrease Propofol Injection Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xingui Dai (Other)
Responsible Party: Sponsor-Investigator, Xingui Dai, MD, First People's Hospital of Chenzhou
Organization: First People's Hospital of Chenzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Warm Decrease Pain
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Injection Site Irritation; Propofol Syndrome; Temperature Change, Body
MeSH Terms: conditions — Propofol Infusion Syndrome; Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: patients for observation will sent to a warmer operating room,while Patients in controled Group will send to normal setting operating room at about 23 centigrade.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not knowing the exact temperature of the room,thought they will have their own feeling about it. Data was collecting with a anesthesia nurse who do not know what will do with these data. data were assessed to an anesthesiologist who did not know the Group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- warmer temperature (Experimental): To compare the incidence and intensity of pain on injection that is caused by propofol in warm temperature（27℃） versus normal temperature(23℃).
  Interventions: Behavioral: warmer temperature
- normal temperature (Placebo Comparator): The purpose of this study is to compare the incidence and intensity of possible pain on injection as well as patient satisfaction caused by propofol in different room temperature(27 VS 23).
  Interventions: Behavioral: warmer temperature

INTERVENTIONS:
Behavioral: warmer temperature — Patients before general anesthesia induction will send to warmer operation Injection pain was accessed with (Visual analogous scale)VAS.

SUMMARY:
Propofol injection pain will be surfed by up to 70-80 percentage by the Patients who induced by propofol. Temperature of Operating room was set to a certain range in normal clinical practice, which is 22- 26 centigrade. Warm feeling will make skin vassal dilated and more blood will pass through to bring more heat out of our body. It had been reported that a bigger venous vessels will get less propofol injection pain.

The investigators hypothesis that Patients who stayed in a warmer room temperature will surf less injection pain while compare to a normal setting room temperature.

ELIGIBILITY:
Inclusion Criteria:

* ASA I~III, aged 18，scheduled or emergency surgery with general anesthesia.

Exclusion Criteria:

* a history of allergy to propofol, allergy to soybean oil
* with peripheral blood diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-28 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
intensity of injection pain | 3 months
  intensity of injection pain was reported by patient themselves before loss their awareness.
numbers of lidocaine rescues for severe injection pain | 3 months
  when unbearable injection happens,patient could ask for stop and 20mg lidocaine was injected as rescue treatments.
incidences of injection pain | 3 months
  Numeric Visual Analog Scale of injection >2 was counted as injection pain happens,the total incidence of injection was compared in two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Chenzhou No.1 People's hopital, Chenzhou, Hunan, China